CLINICAL TRIAL: NCT03769298
Title: Conversion From Immediate Release Tacrolimus to Envarsus XR® in Simultaneous Pancreas-Kidney Recipients: Assessment of Functional, Safety and Quality of Life Outcomes (CIRTEN SPK)
Brief Title: CIRTEN-Simultaneous Pancreas-Kidney Transplant Recipients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0821; A539742 (Other: UW Madison); SMPH/SURGERY/TRANSPLANT (Other: UW Madison); Protocol Version 3/10/2025 (Other: UW Madison)
Record Dates: First submitted 2018-11-16; First posted 2018-12-07 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Kidney Pancreas Transplantation
Keywords: Tremors
MeSH Terms: conditions — Tremor | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: This is a Phase II/III, Single-center, Prospective, Open-label, Single Arm Study of 20 Simultaneous Kidney Pancreas recipients who received a transplant at least 3 months, but no more than 2 years prior, with a history of tremors following transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Envarsus XR (Experimental): Envarsus XR (extended release) will be administered orally, once-daily, for 6 months.
  Interventions: Drug: Envarsus XR

INTERVENTIONS:
Drug: Envarsus XR — The Envarsus XR® drug will be administered to study participants once daily, orally. The dosage can be 0.75 mg, 1 mg or 4 mg. The tacrolimus whole blood trough concentrations will be monitored and titrate Envarsus XR® dosage to achieve target whole blood trough concentration.
  Other Names: tacrolimus

SUMMARY:
This is a Phase II/III, Single-center, Prospective, Open-label, Single Arm Study of 20 Simultaneous Kidney Pancreas recipients who received a transplant at least 3 months, but no more than 5 years prior, with a history of tremors following transplantation.

DETAILED DESCRIPTION:
Accrual objective: Enrollment of 2-3 participants per month and all participants within an 18 month period. With minimum of 1 year follow-up post-conversion, we anticipate the entire study would be completed within 2 ½ years.

Study design: This is a Phase II/III, Single-center, Prospective, Open-label, Single Arm Study of 20 Simultaneous Kidney Pancreas recipients who received a transplant at least 3 months, but no more than 5 years prior, with a history of tremors following transplantation.

Study duration: There will be a minimum of 1 year follow-up post-conversion, and it is expected that the entire study would be completed within 2 ½ years.

Study aims:

* Determine if EnvarsusXR® reduces tremor severity compared to IR tacrolimus
* Determine if EnvarsusXR® improves renal function or glycemic control compared to IR tacrolimus
* Compare the efficacy of EnvarsusXR® by comparing the outcomes (patient, pancreas graft and kidney graft survival) of patients treated with Envarsus XR to those of contemporary and historical controls at our center treated with IR tacrolimus, with the goal of showing non-inferiority.
* Compare insulin resistance and insulin sensitivity by defined measures post conversion between T1D and T2D recipients.

Primary Endpoint:

1. Improvement in patient and physician-assessed degree of tremors based on FTM (Fahn-Tolosa-Martin Tremor Rating Scale) and QUEST (Quality of Life in Essential Tremor Questionnaire) scoring tools
2. Scores on Quality of Life in Essential Tremor and Modified Transplant Symptom Occurrence and Symptom Distress Scale (MTSOSD) Questionnaires

Secondary Endpoints:

1. Renal function - eGFR (estimated glomerular filtration rate) and serum creatinine
2. Glycemic control - AUC by MMTT, fasting BG, fasting C-peptide, calculated C-peptide/glucose ratio, calculated 20/(fasting Cpeptide x fasting BG) as a measure of insulin resistance, calculated HOMA-IR (fasting insulin x fasting BG)/22.5 as a measure of insulin sensitivity/resistance, calculated BETA-2 score to sensitive estimate beta cell function, and HbA1c.
3. Tacrolimus and Mycophenolate doses as well as TAC and MPA levels

ELIGIBILITY:
Inclusion Criteria:

* Adult, 18-70 years of age
* Participant must be able to understand and provide consent
* History of Diabetes Type 1 or Insulin-Dependent Diabetes Type 2 with Chronic Kidney Disease (CKD)
* Recipient of a Simultaneous Pancreas Kidney (SPK) transplant, 3- 60 months prior to screening, per Principal Investigator's discretion.
* Have a history of tremors following transplantation
* Stable pancreas allograft function as evidenced by no requirement of exogenous insulin or oral anti-diabetic agents and stable pancreatic enzymes
* Stable kidney allograft function
* Currently taking Immediate-Release (IR) tacrolimus
* Women of child-bearing potential (WOCP) must have a negative pregnancy test at the time of study entry

Exclusion Criteria:

* Currently maintained on an extended-release tacrolimus immunosuppressive regimen
* Previous history of tremors prior to transplantation
* Solitary pancreas transplant recipients
* History of solid organ transplant other than a kidney or pancreas
* Uncontrolled concomitant infection at the discretion of the investigator
* Presence of Donor Specific Antibodies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in patient and physician-assessed degree of tremors based on Fahn-Tolosa-Marin Tremor Rating Scale | Over 6 months
  FTM-TRS will be used as a tool for essential tremor scoring. (0: no tremor, 1: barely perceptible tremor, 2: < 2 cm, 3: 2-4 cm, and 4: > 4 cm).
Change in patient and physician-assessed degree of tremors based on Quality of Life in Essential Tremor (QUEST) Questionnaire | Over 6 months
  QUEST Questionnaire, a scoring tool will be used to measure the quality of life among patients with Essential Tremor. It consists of 30 items which are rated on a five-point scale (score 0-4), corresponding to the frequency (never, rarely, sometimes, frequently, always) with which tremor was perceived to affect a function or to be associated with various feelings and attitudes. A few items (e.g. 'I had to quit my job because of tremor') could only be answered at the extremes (yes/no; true/false), and these were scored either 0 or 4.
Scores on Quality of Life in Essential Tremor Questionnaires | Over 6 months
  Use QUEST (Quality of Life in Essential Tremor Questionnaire) scoring tool
Scores on Modified Transplant Symptom Occurrence and Symptom Distress Scale (MTSOSD) Questionnaire | Over 6 months
  MTSOSD Questionnaire scores will be used to assess the presence and distress of side effects associated with the use of immunosuppressive drugs after transplantation.

SECONDARY OUTCOMES:
Renal function by eGFR (estimated Glomerular Filtration Rate) | Over 6 months
  Change between baseline and post-conversion as measured by eGFR
Renal function by serum creatinine | Over 6 months
  Change between baseline and post-conversion as measured by serum creatinine
Comparable or improved glycemic control as measured by mixed meal tolerance test | Over 6 months
  Change between baseline and post-conversion
Comparable or improved glycemic control as measured by HbA1c | Over 6 months
  Change between baseline and post-conversion
Tacrolimus doses and levels | Over 6 months
  Change between baseline and post-conversion
Mycophenolate doses and levels | Over 6 months
  Change between baseline and post-conversion

CONTACTS AND LOCATIONS:
Overall Officials: Jon S Odorico, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langone A, Steinberg SM, Gedaly R, Chan LK, Shah T, Sethi KD, Nigro V, Morgan JC; STRATO Investigators. Switching STudy of Kidney TRansplant PAtients with Tremor to LCP-TacrO (STRATO): an open-label, multicenter, prospective phase 3b study. Clin Transplant. 2015 Sep;29(9):796-805. doi: 10.1111/ctr.12581. Epub 2015 Aug 6. PMID 26113208
- [Background] Baraldo M. Meltdose Tacrolimus Pharmacokinetics. Transplant Proc. 2016 Mar;48(2):420-3. doi: 10.1016/j.transproceed.2016.02.002. PMID 27109969
- [Background] Kerstenetzky L, Descourouez JL, Jorgenson MR, Felix DC, Mandelbrot DA, Redfield RR, Odorico JS. A Single-Center Experience With Tacrolimus LCP (Envarsus XR) in Pancreas Transplant Recipients. Ann Pharmacother. 2018 Apr;52(4):392-396. doi: 10.1177/1060028017749076. Epub 2017 Dec 14. No abstract available. PMID 29241340
- [Background] Stacy MA, Elble RJ, Ondo WG, Wu SC, Hulihan J; TRS study group. Assessment of interrater and intrarater reliability of the Fahn-Tolosa-Marin Tremor Rating Scale in essential tremor. Mov Disord. 2007 Apr 30;22(6):833-8. doi: 10.1002/mds.21412. PMID 17343274
- [Background] Ohkura T, Shiochi H, Fujioka Y, Sumi K, Yamamoto N, Matsuzawa K, Izawa S, Kinoshita H, Ohkura H, Kato M, Taniguchi S, Yamamoto K. 20/(fasting C-peptide x fasting plasma glucose) is a simple and effective index of insulin resistance in patients with type 2 diabetes mellitus: a preliminary report. Cardiovasc Diabetol. 2013 Jan 22;12:21. doi: 10.1186/1475-2840-12-21. PMID 23339473
- [Background] Gutch M, Kumar S, Razi SM, Gupta KK, Gupta A. Assessment of insulin sensitivity/resistance. Indian J Endocrinol Metab. 2015 Jan-Feb;19(1):160-4. doi: 10.4103/2230-8210.146874. PMID 25593845
- [Background] Forbes S, Oram RA, Smith A, Lam A, Olateju T, Imes S, Malcolm AJ, Shapiro AM, Senior PA. Validation of the BETA-2 Score: An Improved Tool to Estimate Beta Cell Function After Clinical Islet Transplantation Using a Single Fasting Blood Sample. Am J Transplant. 2016 Sep;16(9):2704-13. doi: 10.1111/ajt.13807. Epub 2016 Apr 21. PMID 27017888
- See also: U.S. Food and Drug Administration. Drug Approval Package. — https://www.accessdata.fda.gov/drugsatfda_docs/nda/2015/206406Orig1_toc.cfm
- See also: Fahn S, Tolosa E, Marin C. Clinical Rating Scale of Tremor — https://www.researchgate.net/publication/307538277_Clinical_Rating_Scale_for_Tremor
- See also: 5. West-Thielke P, Brennan D, Stevens D. Pharmacokinetics of once-daily Envarsus XR in diabetic vs. non-diabetic kidney transplant recipients: a pooled subgroup analysis. [abstract] Kidney Week. Nov 2016, Chicago IL. — https://www.asn-online.org/education/kidneyweek/archives/